CLINICAL TRIAL: NCT05801601
Title: Evaluating Many Ways of Being, an Innovative Gender-synchronized and Gender-transformative Sexual Health Program
Brief Title: Evaluating the Many Ways of Being Program
Acronym: MWB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: Latin American Youth Center (Unknown); Equimundo:Center for Masculinities and Social Justice (Unknown); Family and Youth Services Bureau (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90AP2693
Record Dates: First submitted 2023-02-23; First posted 2023-04-06 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Sexual Behavior; Unprotected Sex
MeSH Terms: conditions — Sexual Behavior; Unsafe Sex

STUDY DESIGN:
Intervention Model Description: This research project will used an individual randomized controlled trial design in which youth at each intervention site will be randomized 1:1 into the experimental condition (Many Ways of Being) or the comparison condition (a career readiness program).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Many Ways of Being (Experimental): In the experimental arm, Equimundo's Many Ways of Being program will be implemented. Youth will receive eight two-hour sessions or 16 one-hour sessions over four to eight weeks for a total of 14 hours and 40 minutes of programming.
  Interventions: Behavioral: Many Ways of Being, an innovative sexual health promotion program focused on addressing rigid gender norms and promoting healthy relationships
- A career readiness program (Active Comparator): In the comparison arm, a curriculum focused on career readiness will be implemented. Youth will receive eight two-hour sessions or 16 one-hour sessions over four to eight weeks for a total of 14 hours and 40 minutes of programming.
  Interventions: Behavioral: A career readiness program

INTERVENTIONS:
Behavioral: Many Ways of Being, an innovative sexual health promotion program focused on addressing rigid gender norms and promoting healthy relationships — The Many Ways of Being program is a gender-synchronous program informed by Equimundo's existing single-gender Manhood 2.0 and Sisterhood 2.0 programs. The curriculum is designed to shift unequal gender attitudes and behaviors and provide skill-building on maintaining healthy relationships, making healthy and informed decisions around sex, and avoiding risky sexual behaviors.
  Other Names: Many Ways of Being
  Arms: Many Ways of Being
Behavioral: A career readiness program — Youth enrolled in the control condition will receive a career readiness curriculum, either International Youth Foundation's Passport to Success, LAYC's Next Generation program or LAYC's Career Readiness Curriculum, depending on the site and implementation period. These programs equip young people with a range of professional, employment readiness, and practical skills that will help them stay in school and acquire the education, professional skills, employment
  Arms: A career readiness program

SUMMARY:
The goal of this randomized control trial is to clinical trial is to evaluate Many Ways of Being, an innovative sexual health promotion program focused on addressing rigid gender norms and promoting healthy relationships.

The overall goal of the MWB program is to reduce incidence of sexually transmitted infections (STI) and unplanned pregnancy and promote healthy, consensual, and violence-free relationships among youth. The primary research question we aim to answer through this study is: Among youth ages 15-19, does the Many Ways of Being program reduce unprotected sex (through consistent and correct use of condoms and contraceptives) compared to the a career readiness program, which does not include sexual health components?

As part of the study, participants will be asked to:

* Attend approximately 14 hours and 40 minutes of programming completed over 4-8 weeks
* Complete baseline, post-intervention, and 9-month follow-up surveys
* For select participants who received the MWB program, participate in an optional focus group discussion

The local evaluation will focus on the impact of the entire MWB intervention, as compared to a similar-length control program focused on career readiness.

ELIGIBILITY:
Inclusion Criteria:

* Youth age 15-19 in the greater Metropolitan DC area

Exclusion Criteria:

* Youth who are actively planning a pregnancy, have participated in the other sexual health programming through the LAYC previously, or are receiving other sexual health education during the implementation period. Youth who do not speak English and/or Spanish will also not be eligible to participate.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Condomless sex (measure 1) | 9 months following program completion
  Vaginal or anal sex without a condom in the past 3 months (yes/no). Yes if had vaginal or anal sex in the past 3 months and did not use a condom "all the time". No if did not have sex or used a condom "all the time".
Unprotected vaginal sex (measure 2) | 9 months following program completion
  Vaginal sex without any contraception (including condom) in the past 3 months (yes/no) Yes if had sex in the past 3 months and did not use a contraceptive "all the time". No if did not have sex or used a contraceptive "all the time".

SECONDARY OUTCOMES:
Sexual agency | 9 months following program completion
  The respondent reported that they communicated what they "liked, disliked, or wanted to try" "all" or "most" of the time and that they asked what their partner "liked, disliked, or wanted to try" "all" or "most" of the time when participating in any sexual activity (including sexual touching) in the past 3 months OR respondent was not sexually active in the past 3 months. (yes/no)
Knowledge related to healthy relationships | Immediately post-program and 9 months following program completion
  Able to identify healthy and unhealthy relationship scenarios (% correct out of 7 items)
Knowledge related to sexual and reproductive health (measure 1) | Immediately post-program and 9 months following program completion
  Knowledge of contraceptive methods (% correct out of 4 items)
Knowledge related to sexual and reproductive health (measure 2) | Immediately post-program and 9 months following program completion
  Knowledge of STIs (% correct out of 5 items)
Knowledge related to sexual and reproductive health (measure 3) | Immediately post-program and 9 months following program completion
  Able to identify sexual consent (% correct out of 4 items)
Intentions to practice sexual health promoting behaviors (measure 1) | Immediately post-program and 9 months following program completion
  Intends to use contraception ("Yes, definitely") if chooses to have sex in the future
Intentions to practice sexual health promoting behaviors (measure 2) | Immediately post-program and 9 months following program completion
  Intends to use condoms ("Yes, definitely") if chooses to have sex in the future
Intentions to practice sexual health promoting behaviors (measure 3) | Immediately post-program and 9 months following program completion
  Intends to visit a health care provider for SRH services in the next 12 months (yes/no "Yes, definitely" vs other responses)
Self-efficacy to practice sexual health promoting behaviors (measure 1) | Immediately post-program and 9 months following program completion
  Know where to go to get birth control (yes/no "Yes, definitely" vs other responses)
Self-efficacy to practice sexual health promoting behaviors (measure 2) | Immediately post-program and 9 months following program completion
  Know where to go to get STI testing/ treatment (yes/no "Yes, definitely" versus other responses)
Self-efficacy to practice sexual health promoting behaviors (measure 3) | Immediately post-program and 9 months following program completion
  Level of comfort going to a provider for services or approaching a trusted adult for information about SRH (4-item Likert scale).
Self-efficacy to practice sexual health promoting behaviors (measure 4) | Immediately post-program and 9 months following program completion
  Self-reported ability to communicate with partners about consent, sex, and contraception (5-item Likert scale). Three items draw from Upadhyay UD et al. Development and Validation of the Sexual and Reproductive Empowerment Scale for Adolescents and Young Adults. J Adolesc Health. 2021 Jan;68(1):86-94.
Positive attitudes around gender | Immediately post-program and 9 months following program completion
  Gender-equitable attitudes scale (7-item Likert scale)
Positive attitudes around sexual health (measure 1) | Immediately post-program and 9 months following program completion
  Self-love subscale from Sexual and Reproductive Empowerment Scale (4-item Likert scale). Citation: Upadhyay UD et al. Development and Validation of the Sexual and Reproductive Empowerment Scale for Adolescents and Young Adults. J Adolesc Health. 2021 Jan;68(1):86-94.
Positive attitudes around sexual health (measure 2) | Immediately post-program and 9 months following program completion
  Sexual pleasure subscale from Sexual Reproductive Empowerment Scale (3-item Likert scale). Citation: Upadhyay UD et al. Development and Validation of the Sexual and Reproductive Empowerment Scale for Adolescents and Young Adults. J Adolesc Health. 2021 Jan;68(1):86-94.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Manlove, PhD, Principal Investigator — Child Trends
Locations (1):
- LAYC's Teen Center, Washington D.C., District of Columbia, United States